CLINICAL TRIAL: NCT03941665
Title: Double Blind Study - Use of Gelronate Gel vs. Aloevera in Preventing/Minimizing Radiation-induced Dermatitis in Breast Cancer Patients
Brief Title: Use of Gelronate Gel vs. Aloevera in Preventing/Minimizing Radiation-induced Dermatitis in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5652-18-SMC
Record Dates: First submitted 2019-05-02; First posted 2019-05-08 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2019-12

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Intervention Model Description: Double blind study
Who Masked: Participant, Investigator
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gelronate (Experimental): Tested new medical device
  Interventions: Device: Gelronate; Other: Aloevera
- Aloevera (Active Comparator): Current product used by the medical center
  Interventions: Device: Gelronate; Other: Aloevera

INTERVENTIONS:
Device: Gelronate — Gel for topical use
Other: Aloevera — Gel for topical use

SUMMARY:
The aim of the study is to evaluate the effect of Gelronate gel, NaHA based product (medical device for topical application) vs. Aloevera gel, in prevention or minimizing of radiation induced skin reaction in breast cancer patients

DETAILED DESCRIPTION:
Gelronate is gel composed of 1% high molecular weight pharmaceutical grade sodium hyaluronate and preservatives dissolved in pharmaceutical grade purified water. Gelronate supply in an airless pump bottle contain ~30 ml gel. In the study, 120 female patients planned to receive whole breast radiation (with or without lymphatic drainage) in the radiotherapy unit at Sheba Medical Center.

Patients will undergo CT simulation with 3D treatment planning (as routine done) and will receive 42.4 Gy in daily fraction of 2.65 Gy, five times per week to the whole breast according to the standard department protocol, with or without concomitant or subsequent lumpectomy cavity boost. Patients data including demographics, staging, systemic therapy, radiation details, other medications will be recorded the protocol's forms.

The gel will be applied as a thin lotion twice a day, immediately after radiotherapy treatment and once more in the evening/morning. The therapy will continue for 10 days following the end of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged at least 18 years with unilateral breast following lumpectomy +/- chemotherapy
* Planned to receive 42.4 Gy whole breast irradiation +/- boost to tumor bed.
* ECOG performance status 0-2.
* Capable of giving written informed consent.
* No co-morbidities known to affect radiotherapy reactions.
* No co-existing acute or chronic skin disease.
* No evidence of infection or inflammation of breast to be treated.
* Not receiving chemotherapy during radiotherapy course. Biological therapy (e.g. Herceptin) or hormone therapy will be allowed during the study.

Exclusion Criteria:

* Chemotherapy within 4 weeks prior to planned start of radiation or chemotherapy planned during radiation.
* Prior radiotherapy to the chest wall.
* Collagen vascular disease.
* Participation in other clinical study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
Development and degree of any skin reaction | 4 weeks
  Grading according to Radiation Toxicity Grading (RTOG) skin toxicity score. Full scale of RTOG is 0 (no change over baseline) to 4 (ulceration, hemorrhage, necrosis).
Development and degree of any skin reaction | 4 weeks
  Assessment of skin reaction by scoring of weekly digital photographs
Development and degree of any skin reaction | 4 weeks
  Patient comfort assessed by weekly administrated questionnaire. Scores are between 1 (nothing) to 4 (all over the breast)

SECONDARY OUTCOMES:
Skin reaction requiring conventional topical therapy | 4 weeks
  Skin reaction requiring conventional topical therapy (e.g. steroid cream etc.) as evaluated by clinical. judgment of radiotherapy nurse/radiation oncologist at OTV (on treatment view visit that will include RTOG (Radiation Toxicity Grading) scores (in the range 0 no change to 4 ulceration, hemorrhage, necrosis) and dermatology assessment according to the table in the protocol (general view range 1 (nothing) to 4 (continuous))

CONTACTS AND LOCATIONS:
Overall Officials: Ofer S Dubinsky, Ph.D., Study Director — Ferring Holding Ltd.
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Primavera G, Carrera M, Berardesca E, Pinnaro P, Messina M, Arcangeli G. A double-blind, vehicle-controlled clinical study to evaluate the efficacy of MAS065D (XClair), a hyaluronic acid-based formulation, in the management of radiation-induced dermatitis. Cutan Ocul Toxicol. 2006;25(3):165-71. doi: 10.1080/15569520600860009. PMID 16980242
- [Result] Leonardi MC, Gariboldi S, Ivaldi GB, Ferrari A, Serafini F, Didier F, Mariani L, Castiglioni S, Orecchia R. A double-blind, randomised, vehicle-controlled clinical study to evaluate the efficacy of MAS065D in limiting the effects of radiation on the skin: interim analysis. Eur J Dermatol. 2008 May-Jun;18(3):317-21. doi: 10.1684/ejd.2008.0396. Epub 2008 May 13. PMID 18474463

DOCUMENTS (1):
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT03941665/Prot_000.pdf